CLINICAL TRIAL: NCT02260609
Title: A Multicenter, Open-label, Single-Arm Study to Evaluate the Safety and Efficacy of GrafixCORE® for the Treatment of Complex Diabetic Foot Wounds With Exposed Tendon and/or Bone
Brief Title: GrafixCORE®: Open-Label Study to Evaluate the Safety and Efficacy of GrafixCORE® for Complex Diabetic Foot Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osiris Protocol 310
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Complex Diabetic Foot Wounds
Keywords: Complex Wound; Diabetic Foot Ulcer; DFU; GrafixCORE; Exposed tendon; Exposed bone; Allograft tissue
MeSH Terms: conditions — Diabetic Foot | interventions — Histocompatibility Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label (Other): Grafix®: Cryopreserved Placental Membrane
  Interventions: Other: Grafix®

INTERVENTIONS:
Other: Grafix® — The treatment indication is for complex diabetic foot wounds with exposed tendon and/or bone that can accommodate up to three 5cm x 5cm pieces of Grafix®.
  Patients will be treated for up to 16 weeks.
  Patients will be evaluated at screening and then weekly throughout the study or until wound closure.
  Other Names: Tissue; Allograft Tissue

SUMMARY:
A multicenter, open-label, single-arm study to evaluate the safety and efficacy of GrafixCORE® for the treatment of complex diabetic foot wounds with exposed tendon and/or bone.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years and 85 years of age inclusive, as of the date of screening
2. Confirmed diagnosis of Type I or Type II Diabetes
3. Index wound graded in the Texas Classification System as Grade II-III, Stage A or C (without active infection)
4. Wound is located on the foot below the malleoli
5. Wound accommodates up to three (3) 5 cm x 5 cm pieces of GrafixCORE® that completely cover the wound
6. Patient's wound extends through the dermis and into subcutaneous tissue with evidence of exposed muscle, tendon, bone, and/or joint capsule
7. Patient has adequate circulation to the foot as documented by either:

   * Ankle Brachial Index (ABI) ≥ 0.5 and ≤ 1.2, or
   * In patients with non-compressible ankle vessels, a Toe BP ≥ 40 mmHg or TcPO2 > 30 mmHg, or
   * Skin perfusion pressure > 30 mmHg

Exclusion Criteria:

1. Index Wound is of non-diabetic pathophysiology
2. Gangrene is present on any part of the affected foot
3. Index Wound is over a Charcot deformity
4. The longest dimension of the Index Wound exceeds 15 cm at the Baseline Visit
5. Patient has a glycated hemoglobin A1 (HbA1c) level of >14%
6. Requiring intravenous (IV) antibiotics to treat the index wound infection at enrollment
7. Patient has a wound within 15cm of the Index Ulcer identified for study consideration
8. Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents
9. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
10. Current evidence of osteomyelitis, cellulitis, or other evidence of infection including fever or pus drainage from the wound site
11. Patient has active malignancy other than non-melanoma skin cancer
12. Patient's random blood sugar is >450 mg/dl at screening
13. Patient has untreated alcohol or substance abuse at the time of screening, or is deemed to be non-adherent to the protocol by the Investigator
14. Pregnant women
15. Patient is currently enrolled or participated in another investigational device, drug, or biological trial within 30 days of screening
16. Patient has allergy to primary or secondary dressing materials used in this trial
17. Patient has had within the last 14 days, or is currently undergoing, or is planning for wound treatments with enzymes, growth factors, living skin, dermal substitutes or other advanced biological therapies
18. In the opinion of the Investigator, the patient is unsuitable for participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
100% granulation of wound as determined by the investigator | Up to 16 weeks after the Initial Treatment Visit

SECONDARY OUTCOMES:
Time to 100% granulation | Up to 16 weeks after the Initial Treatment Visit
Number of applications of Grafix® | Up to 16 weeks after the Initial Treatment Visit
Measurement of percent wound area reduction as determined by the investigator | Up to 16 weeks after the Initial Treatment Visit
Closure of wound defined by 100% re-epithelialization | Up to 16 weeks after the Initial Treatment Visit

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Carl T. Hayden Medical Research Foundation, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Miami VA, Miami, Florida
  - South Shore Hospital, Weymouth, Massachusetts